CLINICAL TRIAL: NCT01709630
Title: Pharmacokinetics (PK)/Pharmacodynamics (PD) Modeling of Magnesium Sulfate In the Mother and Exposed Neonate
Brief Title: PK/PD Modeling of Magnesium in the Mother and Neonate
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Associate Professor, Stanford University
Other Study IDs: ID-2803
Record Dates: First submitted 2012-10-14; First posted 2012-10-18 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Magnesium Sulfate Pharmacokinetics and Pharmacodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimens will be obtained to test magnesium levels in the mother and neonate.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neonatal: Neonates born to pregnant women exposed to magnesium sulfate for preeclampsia, tocolysis, or neuroprotection.
  Interventions: Drug: Magnesium sulfate infusion
- Maternal: Pregnant women exposed to magnesium sulfate for preeclampsia, tocolysis, or neuroprotection
  Interventions: Drug: Magnesium sulfate infusion

INTERVENTIONS:
Drug: Magnesium sulfate infusion — Participants will be given magnesium sulfate infusion as part of their normal care for either preeclampsia, tocolysis, or neuroprotection.

SUMMARY:
Determine significant correlations between maternal serum magnesium levels, and maternal and neonatal outcomes.

DETAILED DESCRIPTION:
We will construct a pharmacokinetic and pharmacodynamic model of intravenous magnesium sulfate administered antenatally to expectant mothers and exposed fetuses with the aim of optimizing maternal and fetal outcomes while preventing maternal and neonatal overdosing and morbidity associated with current magnesium treatment protocols. Once we have developed a PK/PD model in our own hospital cohort, we will apply this model to a large existing NICHD database to mathematically calculate optimal dosing protocols.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18-45 years
* Magnesium sulfate exposure for preeclampsia, tocolysis, or neuroprotection
* Neonates (male or female) born at 24-42 weeks gestation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and neonates exposed to magnesium sulfate infusion around the time of delivery for one of three reasons: 1.) preeclampsia 2.) tocolysis 3.) neuroprotection.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maternal and neonatal blood magnesium levels | 24 months
  Pregnant women and neonates exposed to magnesium sulfate for preeclampsia, tocolysis, or neuroprotection will have blood samples drawn at set time points around the time of delivery.

SECONDARY OUTCOMES:
Maternal and neonatal side effects | 24 months
  Maternal drug side effects (flushing, sedation, nausea, vomiting, respiratory rate, oxygen saturations, blood pressure, heart rate, and patella tendon reflex depression) will be assessed prospectively.
  Neonatal drug effects: Incidence of cerebral palsy, neonatal mortality, NICU and special care admissions, respiratory distress, intraventricular hemorrhage, necrotizing enterocolitis, hypotonia, feeding difficulties, and diagnosis of hypermagnesemia will be recorded, We will use validated and standardized definitions for diagnoses and all clinical outcome measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital at Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Background] Rouse DJ, Hirtz DG, Thom E, Varner MW, Spong CY, Mercer BM, Iams JD, Wapner RJ, Sorokin Y, Alexander JM, Harper M, Thorp JM Jr, Ramin SM, Malone FD, Carpenter M, Miodovnik M, Moawad A, O'Sullivan MJ, Peaceman AM, Hankins GD, Langer O, Caritis SN, Roberts JM; Eunice Kennedy Shriver NICHD Maternal-Fetal Medicine Units Network. A randomized, controlled trial of magnesium sulfate for the prevention of cerebral palsy. N Engl J Med. 2008 Aug 28;359(9):895-905. doi: 10.1056/NEJMoa0801187. PMID 18753646
- [Background] Pryde PG, Mittendorf R. Contemporary usage of obstetric magnesium sulfate: indication, contraindication, and relevance of dose. Obstet Gynecol. 2009 Sep;114(3):669-673. doi: 10.1097/AOG.0b013e3181b43b0e. PMID 19701048
- [Background] Greenberg MB, Penn AA, Whitaker KR, Kogut EA, El-Sayed YY, Caughey AB, Lyell DJ. Effect of magnesium sulfate exposure on term neonates. J Perinatol. 2013 Mar;33(3):188-93. doi: 10.1038/jp.2012.95. Epub 2012 Jul 26. PMID 22836873